CLINICAL TRIAL: NCT04232111
Title: Effect of AVACEN 100 on Brachial Artery Blood Flow
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never took off and the sponsor lost interest.
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AVACENBF
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Blood Flow

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Thermoneutral (Sham Comparator): Neither heat nor vacuum applied to hand
  Interventions: Device: sham
- Heat and Vacuum (Experimental): Heat and vacuum applied to hand
  Interventions: Device: Heat; Device: Vacuum
- Heat only (Experimental): Only heat applied to hand
  Interventions: Device: Heat

INTERVENTIONS:
Device: Heat — Heat applied to hand
  Arms: Heat and Vacuum; Heat only
Device: Vacuum — vacuum applied to hand
  Arms: Heat and Vacuum
Device: sham — neither heat nor vacuum
  Arms: Thermoneutral

SUMMARY:
Determine effect of AVACEN 100 on brachial artery blood flow

DETAILED DESCRIPTION:
Blood flow measured via ultrasound doppler

ELIGIBILITY:
Inclusion Criteria:

* anyone within specified age

Exclusion Criteria:

* anyone outside specified age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
brachial artery blood flow via ultrasound doppler | 10 min
brachial artery blood flow via ultrasound doppler | 20 min
brachial artery blood flow via ultrasound doppler | 30 min

IPD SHARING:
Plan to Share IPD: No